CLINICAL TRIAL: NCT02454283
Title: RESTORE SR: A Multi-center, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of a Single Oral Dose of Vanoxerine for The Conversion Of Subjects With REcent Onset Atrial Fibrillation or Flutter to Normal Sinus Rhythm
Brief Title: Safety and Efficacy of Vanoxerine for the Conversion of Subjects With Recent Onset Atrial Fibrillation or Flutter to Normal Sinus Rhythm
Acronym: RESTORE SR
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Cardiac safety finding
Sponsor: Laguna Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LGN-VN-003
Record Dates: First submitted 2015-05-20; First posted 2015-05-27 (Estimated); Results first posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-06

CONDITIONS: Atrial Fibrillation or Flutter
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vanoxerine HCl (Experimental): Vanoxerine HCl, 400 mg (2 x 200 mg capsules), orally, single dose
  Interventions: Drug: Vanoxerine HCl
- Placebo (Placebo Comparator): identically matching placebo capsules, orally, single-dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vanoxerine HCl
  Arms: Vanoxerine HCl
Drug: Placebo
  Arms: Placebo

SUMMARY:
LGN-VN-003 is a prospective, multi-center, randomized, double-blind, placebo-controlled study to evaluate the safety and efficacy of a single oral dose of vanoxerine for the conversion of subjects with recent onset atrial fibrillation (AF) or atrial flutter (AFL) to normal sinus rhythm. Up to 625 subjects will be randomized in a 2:1 fashion so at least 400 vanoxerine and 200 placebo subjects receive study drug.

ELIGIBILITY:
Inclusion Criteria:

* Subject has been informed of the investigational nature of this study and has given written informed consent in accordance with institutional, local, and national guidelines.
* Able to return for Day 8 follow up.
* Male or female 18 years of age or greater.
* Onset of AF/AFL within the 7 calendar days preceding randomization, based on symptoms.
* AF/AFL documented by ECG during the screening period.
* Adherence to local clinical standards or the ACC/AHA or ESC practice guidelines for AF/AFL regarding thromboembolic event prevention and treatment.

Exclusion Criteria:

* Previous exposure to vanoxerine HCl.
* Women of childbearing potential (neither surgically sterilized nor post-menopausal defined as cessation of menses for over one year)
* Systolic blood pressure <110 mmHg (unless documented to be usual value).
* Average heart rate <60 bpm documented by screening ECG.
* Average QTc >440 msec documented by screening ECG.
* QRS interval >140 msec documented by screening ECG.
* Paced atrial rhythm on screening ECG.
* History of receiving another Class I or Class III antiarrhythmic drug within 3 days prior to randomization. Excluded Class I antiarrhythmic drugs include quinidine, procainamide, disopyramide, lignocaine, mexilitine, flecainide, and propafenone. Excluded Class III drugs include dofetilide, sotalol, dronedarone, and ranolazine.
* History of amiodarone (oral or IV) within the 90 days prior to randomization.
* Native or prosthetic aortic or mitral stenosis with aortic valve area ≤1.0 cm2 or mitral valve area of <1.5 cm2 or any other valvular diseases for which surgery is indicated.
* Treatment with any loop diuretic (e.g., furosemide, bumetanide, torsemide, ethacrynic acid, etc.) in the 30 days prior to randomization.
* Ejection fraction of <35% within the 3 months prior to randomization (most recent measure if more than one).
* AF/AFL as a result of surgery (postoperative AF/AFL) within 30 days prior to randomization.
* History of electrical cardioversion within the 7 calendar days prior to randomization.
* History of any polymorphic ventricular tachycardia including torsades de pointes.
* History or family history of long QT syndrome or other inherited arrhythmia syndrome.
* History of ventricular tachycardia requiring drug or device therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (4):
  - Littleton, Colorado
  - Washington D.C., District of Columbia
  - Iowa City, Iowa
  - St Louis, Missouri
- Bulgaria (2):
  - Plovdiv
  - Sofia
- Hungary (5):
  - Budapest
  - Hódmezővásárhely
  - Pécs
  - Rókus
  - Zalaegerszeg
- Israel (2):
  - Ashkelon
  - Safed
- Russia (3):
  - Moscow
  - Saint Petersburg
  - Vladimir

RESULTS

PARTICIPANT FLOW:
Groups:
- Vanoxerine HCl: Vanoxerine HCl, 400 mg (2 x 200 mg capsules), orally, single dose
  Vanoxerine HCl
- Placebo: identically matching placebo capsules, orally, single-dose
  Placebo
Period: Overall Study
Arm/Group | Vanoxerine HCl | Placebo
Started | 26 | 15
Completed | 26 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vanoxerine HCl | Placebo | Total
Number analyzed (Participants) | 26 | 15 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (9.3) | 66.9 (11.3) | 67.7 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 21 | 8 | 29
Prior AF/AFL [Number; unit: participants] | 16 | 7 | 23
Hypertension [Number; unit: participants] | 16 | 11 | 27
Diabetes mellitus [Number; unit: participants] | 4 | 0 | 4
Hyperlipidemia [Number; unit: participants] | 8 | 6 | 14
COPD [Number; unit: participants] | 2 | 1 | 3
Hyperthyroidism [Number; unit: participants] | 1 | 0 | 1
Hypothyroidism [Number; unit: participants] | 3 | 0 | 3
Prior stroke [Number; unit: participants] | 0 | 2 | 2
Pacemaker [Number; unit: participants] | 1 | 0 | 1
Heart failure [Number; unit: participants] | 5 | 2 | 7
LVEF, mean [Mean (Standard Deviation); unit: %] | 54.3 (8.4) | 55.1 (12.4) | 54.6 (9.7)
Mitral stenosis [Number; unit: participants] | 0 | 0 | 0
Mitral regurgitation [Number; unit: participants] | 10 | 4 | 14
Aortic stenosis [Number; unit: participants] | 1 | 0 | 1
Aortic regurgitation [Number; unit: participants] | 4 | 1 | 5
Ischemic heart disease [Number; unit: participants] | 3 | 3 | 6
Prior revascularization (PCI or CABG) [Number; unit: participants] | 2 | 2 | 4
Prior antiarrhythmic drug therapy [Number; unit: participants] | 0 | 2 | 2
Prior catheter ablation of AF [Number; unit: participants] | 1 | 0 | 1
Aspirin [Number; unit: participants] | 5 | 2 | 7
Warfarin [Number; unit: participants] | 3 | 1 | 4
Non vitamin K antagonist [Number; unit: participants] | 4 | 2 | 6
Other anticoagulant [Number; unit: participants] | 11 | 3 | 14

OUTCOME MEASURES:

1. Primary Outcome: Conversion to Sinus Rhythm
Description: Conversion to sinus rhythm (or atrial paced rhythm in the case of subjects with a pacemaker and atrial leads) documented by ECG (Holter ECG, 12-lead ECG, monitor lead ECG, or other format ECG) of at least 1 continuous minute within the 24 hours defined by the time of study drug administration through 24 hours after the time of study drug administration.
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Vanoxerine HCl | Placebo
Number analyzed (Participants) | 26 | 15
participants | 18 | 3

2. Secondary Outcome: Length of Stay (From Time of Study Drug Administration)
Time Frame: 8 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Vanoxerine HCl | Placebo
Number analyzed (Participants) | 20 | 12
days | 4.7 (3.2) | 4.2 (2.9)

ADVERSE EVENTS:
Arm/Group | Vanoxerine HCl | Placebo
Serious Adverse Events (participants affected / at risk) | 4/26 | 0/15
Other Adverse Events (participants affected / at risk) | 0/26 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vanoxerine HCl (N=26) | Placebo (N=15)
polymorphic ventricular tachycardia (Cardiac disorders) | 3 (3) | 0 (0)
torsades de pointes (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No